CLINICAL TRIAL: NCT04483063
Title: Can Additional Preoperative Skin Cleaning on Face, Neck and Chest With Chlorhexidine Reduce Cutibacterium Acnes Contamination on Sutures in Arthroscopy Rotator Cuff Repair?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Kai-Lan Hsu, Attending physician, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-BR-108-052
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: C. Acnes; Arthroscopic Rotator Cuff Repair

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extended shoulder group (Experimental): 2% chlorhexidine gluconate skin cleanser over the not only the operative shoulder and axilla but also the chest, back, neck, and face
  Interventions: Drug: 2% chlorhexidine gluconate skin cleanser
- Shoulder group (Experimental): 2% chlorhexidine gluconate skin cleanser over the operative shoulder and axilla
  Interventions: Drug: 2% chlorhexidine gluconate skin cleanser
- Control group (No Intervention): Skin prepare with soap as usual

INTERVENTIONS:
Drug: 2% chlorhexidine gluconate skin cleanser — 2% chlorhexidine gluconate skin cleanser over shoulder region before shoulder surgery
  Arms: Extended shoulder group; Shoulder group

SUMMARY:
The purpose of our study was to investigate whether preoperative skin cleaning on face, neck, and chest with chlorhexidine could reduce suture contamination of C. acnes in arthroscopic rotator cuff repair. We hypothesized that preoperative skin cleaning on face, neck and chest with chlorhexidine can reduce C. acnes contamination on sutures in arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* primary arthroscopic rotator cuff repair

Exclusion Criteria:

* younger than 18 years
* having previous shoulder surgeries or shoulder infection episodes
* having a history of allergy to chlorhexidine
* who refused to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Culture positive | Within 2 weeks postoperatively
  Culture positive for C. acnes from the suture used in the arthroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No